CLINICAL TRIAL: NCT07189390
Title: A Randomised Controlled Trial to Assess if a Probiotic Intervention Leads to Enhanced Immune Responses to Vaccination in Antibiotic-treated Infants (Bloom Infant Probiotic (BIP) Study)
Brief Title: The Bloom Infant Probiotic (BIP) Study
Acronym: BIP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: South Australian Health and Medical Research Institute (Other)
Collaborators: Flinders University (Other); Women's and Children's Hospital, Adelaide (Unknown); Flinders Medical Center (Unknown); Women's & Children's Hospital Foundation (Unknown); The University of Western Australia (Other)
Responsible Party: Principal Investigator, David Lynn, Professor, South Australian Health and Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025/HRE00173
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Infant, Newborn; Immunity; Immunisation; Antibiotic Treatment; Microbiome Dysbiosis
Keywords: infant; newborn; neonate; antibiotic; microbiome; microbiota; gut; probiotics; bifidobacteria; bifidobacterium; infloran; immunisation; immunity; immune system; vaccine; vaccination; immunization; randomised controlled trial; randomized controlled trial
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): These participants will receive a probiotic, daily for fourteen days.
  Interventions: Drug: Probiotic
- Control (Placebo Comparator): These participants will receive a placebo (contains the same excipients as the probiotic but no bacterial strains), daily for fourteen days.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Probiotic — Probiotic capsule contents will be dissolved in a small amount of breast milk, formula or sterile water (drinking water boiled, then cooled) and administered by the infant's parent/guardian to infants as an oral bolus dose. Probiotic Infloran® Hard capsules (Bifidobacterium bifidum & Lactobacillus acidophilus) are a listed medicine on the Australian Register of Therapeutic Goods (ARTG). Infloran® has been previously used in infants including pre-term infants for other indications including supporting healthy digestion or improving digestive system flora. Infloran® is manufactured by Laboratorio Farmaceutico SIT S.r.l., Via Cavour 70 - 27035 Mede (PV) Italy.
  Other Names: Infloran®
  Arms: Probiotic
Drug: Matching placebo — Placebo contains the same excipients as Infloran, it is also made from the same capsule, but it does not contain any bacterial strains. Placebo capsule contents will be dissolved in a small amount of breast milk, formula or sterile water (drinking water boiled, then cooled) and administered by the infant's parent/guardian to infants as an oral bolus dose. The placebo is manufactured by Syntro Health, 558-562 Swan St, Richmond, VIC 3121.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to investigate whether administering a probiotic (Infloran®) to infants who received antibiotics in the first 28 days of life can restore or enhance their immune response to routine vaccines.

Antibiotic use in the first weeks of life can lower the levels of beneficial gut bacteria, such as bifidobacteria, which play a key role in immune function. As a result, infants treated with antibiotics may produce fewer antibodies after routine vaccinations, leaving them less protected against infections.

The main questions this study aims to answer are:

* Does treatment with the probiotic Infloran® improve the geometric mean concentrations (GMCs) of anticapsular antibodies against at least 11 serotypes included in the pneumococcal conjugate vaccine (PCV20) in serum samples collected at 6 months of age compared with placebo in infants treated with antibiotics in the neonatal period?
* Does treatment with the probiotic Infloran® improve the GMCs for the pneumococcal conjugate vaccine (PCV20) at 12 months of age compared with placebo in infants treated with antibiotics in the neonatal period?
* Does treatment with the probiotic Infloran® improve the GMCs of other routine childhood vaccines at 6 and 12 months of age compared with placebo in infants treated with antibiotics in the neonatal period?
* Does treatment with the probiotic Infloran® increase the proportion of infants achieving seroprotective antibody levels for pneumococcal antigens compared to placebo in infants treated with antibiotics in the neonatal period?
* What are the differences in antigen specific T cell responses, flow cytometry, blood transcriptomics, and gut microbiota composition in the probiotic (Infloran®) vs placebo groups in infants treated with antibiotics in the neonatal period?

Researchers will compare infants who receive Infloran® (a probiotic containing Bifidobacterium bifidum and Lactobacillus acidphilus) with those who receive a placebo (which contains the same excipients as Infloran® but does not contain any bacterial strains).

Participants will:

* Be randomly assigned to receive either a 14-day course of probiotic Infloran® or a placebo.
* Provide blood samples (3-5 mL) at 6 weeks, 6.5 weeks (optional blood-draw for exploratory endpoint), 6 months and 12 months of age.
* Provide stool samples at four timepoints: prior to starting the intervention (probiotic/placebo), on day 7, on day 14 after completion of the study supplement, and prior to their first vaccination at 6 weeks of age.
* Receive routine vaccinations at 6 weeks, 4 months and 6 months in line with the National Immunisation Program
* Complete surveys to collect information regarding probiotic/placebo administration and vaccination related side effects

This study aims to recruit 360 infants to assess whether this probiotic treatment following antibiotic exposure improves the immunogenicity of vaccinations. The information from this study will improve our understanding of how probiotic intervention can support optimal immune responses to vaccination in early life. The findings could potentially influence public health strategies, offering a new way to support optimal vaccine responses in antibiotic-treated infants.

ELIGIBILITY:
Inclusion Criteria:

1. Infants administered antibiotics in the first 28 days of life. Infants must have documented direct antibiotic exposure - defined as having received at least 36 hours of antibiotic treatment in the neonatal period (the first 28 days after birth).
2. Gestational age ≥ 35 weeks.
3. Birth weight ≥ 2500g.
4. Mother aged at least 18 years and able and willing to provide written informed consent for themselves and their infant.
5. Parent/guardian agrees to not give any other probiotics to their infant prior to vaccination at 6 weeks, including any formula that contains probiotics.
6. Infant planning to receive all nationally approved vaccines during next 6 months.

Exclusion Criteria:

1. Significant medical condition in either the mother or infant that, in the opinion of a medical investigator, may interfere with the study.
2. Infant had confirmed sepsis or other serious infection in the neonatal period.
3. Infants with known congenital diseases or who are immunocompromised or considered medically at risk (MAR).
4. Infant participating in another interventional trial during the trial period.

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
The Geometric Mean Concentrations (GMCs) of anticapsular antibodies against at least 11 serotypes included in the pneumococcal conjugate vaccine (PCV20) in serum collected at 6 months in the probiotics vs placebo group. | 6 months

SECONDARY OUTCOMES:
The GMCs for at least 11 serotypes included in pneumococcal conjugate vaccine (PCV20) as measured by serum assay at 12 months in the probiotic vs. placebo group. | 12 months
The GMCs for other vaccine antigens (e.g. diphtheria, tetanus and pertussis toxoids, Haemophilus influenzae type b polyribosylribitol phosphate, Hepatitis B surface antigen) as measured by serum assays at 6 and 12 months in both arms. | 12 months
Proportion of infants achieving seroprotective antibody levels (i.e. seroprotection) for pneumococcal antigens. | 12 months

OTHER OUTCOMES:
Activation-induced markers (AIM) assays will be performed to assess antigen-specific CD4 and CD8 T cell responses in probiotic vs. placebo groups. | 12 months
Flow cytometry analysis of blood samples to compare immune cell frequencies and activation marker expression in probiotic vs. placebo groups. | 12 months
Blood transcriptomics using RNA (ribonucleic acid) sequencing to measure gene expression responses to immunisation (i.e. which genes are turned on or off in blood) in probiotic vs. placebo groups. | Before and after the participants' 6-week immunisations
Assessment of bacterial load (qPCR (quantitative Polymerase Chain Reaction) assay) and microbial composition of the stool microbiota using metagenomics (microbial DNA sequencing) in probiotic vs. placebo groups. | 2 months
Correlative analysis of metagenomic, transcriptomic, and immunological datasets. | 12 months
Assessment of whether probiotic supplementation influences the incidence and severity of respiratory infections during the first 12 months of life. | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Women's and Children's Hospital, Adelaide, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable individual participant data, from participants who give specific consent, may be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept SAHMRI's conditions, under a collaborator agreement, for accessing:
  * Individual participant data that underlie the results reported in our articles after deidentification (text, tables, figures and appendices)
  * Study protocol, Statistical Analysis Plan, PICF
  Molecular data generated from this study (i.e. transcriptomic, epigenomic and metagenomic) will be labelled with a unique identification code and stored on an appropriate data repository (e.g. Gene Expression Omnibus, Sequence Read Archive) with demographic information (age and sex). No identifying participant information will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: At the time of publication. Data will be available indefinitely.
Access Criteria: Researchers from a recognised research institution can approach SAHMRI for access of data. The researcher will need to provide evidence that the proposed use of the data has been ethically reviewed and approved by an Institutional Review Board (IRB)/ Human Research Ethics Committee (HREC), and accept SAHMRI's conditions, under a collaborator agreement.